CLINICAL TRIAL: NCT02127424
Title: Targeted Nurse-driven HIV Screening Using Rapid Tests in Emergency Departments in the Metropolitan Paris Region
Brief Title: Targeted Nurse-driven HIV Screening in Emergency Departments
Acronym: DICI-VIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: K130601
Record Dates: First submitted 2013-12-19; First posted 2014-04-30 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-04

CONDITIONS: Targeted HIV Screening, Emergency Departments
Keywords: Nurse; Nursing; Screening; HIV; Emergency Service Hospital
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination of the nurse-driven HIV targeted screening and the (Experimental): Nurses will offer screening to all patients at EDs, aged 18-64 years old, identified as high-risk by a self-administered questionnaire, not know to be HIV positive, accepting to participate by providing an informed consent and not being seen at ED for post-exposure prophylaxis or unstable medical illness. The questionnaire was previously tested in one ED. In case of reactive rapid test result, blood specimen will be collected for standard enzyme-linked immunosorbent assay and Western blot confirmation. A follow-up visit with an on-site infectious disease specialist will be arranged within the following 48 hours.
  Interventions: Procedure: Nurse-driven HIV targeted screening
- Current practice (no intervention) (Active Comparator): Physician-directed HIV diagnostic testing
  Interventions: Procedure: Current practice

INTERVENTIONS:
Procedure: Nurse-driven HIV targeted screening
  Arms: Combination of the nurse-driven HIV targeted screening and the
Procedure: Current practice
  Arms: Current practice (no intervention)

SUMMARY:
To reduce late HIV diagnosis that remains common in France, the national health agency has promoted non-targeted HIV screening in health care settings, including emergency departments (EDs). In our previous survey, non-targeted nurse-driven HIV screening by rapid tests was feasible, well-accepted but identified only a few new HIV diagnoses mostly among patients at high-risk. Our findings, consistent with results from other international groups, suggest that a targeted strategy could be feasible, efficient and cost-effective with fewer tests required. However, the feasibility and the efficacy of this strategy remain unknown in France.

The main aim of the present study is to compare the efficacy of 2 strategies: 1) the combination of the nurse-driven HIV targeted screening and the current practice (physician-directed HIV diagnostic testing) versus 2) the current practice alone.

The strategies will be compared during 2 randomly assigned periods (cluster randomization and cross-over) in 8 EDs of metropolitan Paris.

During targeted period, nurses will offer screening to all patients at EDs, aged 18-64 years old, identified as high-risk by a self-administered questionnaire, not know to be HIV positive, not being seen for post-exposure prophylaxis or unstable medical illness, and accepting to participate by providing an informed consent.

In case of confirmed reactive rapid test result, a follow-up visit with an on-site infectious disease specialist will be arranged within the following 48 hours.

DETAILED DESCRIPTION:
Background :

Despite easy and free access to HIV testing services and 5 million of tests per year performed, late diagnosis remains common in France with one-third of HIV infections diagnosed associated with AIDS or CD4 lymphocyte counts of less than 200/μL. To improve early detection, the national health agency has promoted non-targeted HIV screening in health care settings, including emergency departments (EDs), in addition to diagnostic testing routinely performed by physicians. In our previous survey conducted in 2009-2010 in 29 EDs of the metropolitan Paris area, non-targeted nurse-driven HIV screening by rapid tests was feasible, well-accepted but identified only a few new HIV diagnoses mostly among patients at high-risk. Our findings, consistent with results from other international groups, suggest that a targeted strategy could be feasible, efficient and cost-effective with fewer tests required. However, the feasibility and the efficacy of this strategy remain unknown in France.

Primary objective :

The aim of the present study is to compare the efficacy of two strategies: 1) the combination of the nurse-driven HIV targeted screening and the current practice (physician-directed HIV diagnostic testing) versus 2) the current practice alone (physician-directed HIV diagnostic testing).

The main outcome measure is the number of patients with newly identified HIV infection among the number of 18-64 years patients visited EDs (apart from being seen for prophylaxis after exposure to HIV) during the inclusion periods.

Secondary objectives :

The linkage into care of patients with newly diagnosed infection, the number of new HIV positive tests among the total number of tests, and the early detection will be compared.

The feasibility of the nurse-driven HIV screening (proportion of : filled-questionnaires, proposition of the nurse-driven HIV screening, acceptation by patients and HIV rapid tests done by nurses) and its acceptability caregivers in each ED will be evaluated as well as its cost-effectiveness.

Methods :

Multicenter trial with cluster randomization and cross-over The 2 strategies will be compared during 2 randomly assigned periods separated by a month (cluster randomization and cross-over). 8 750 patients per ED and per period are expected with 8 EDs (cf. statistical plan).

The study will be performed in 8 EDs of metropolitan Paris, an area in which half of France's new HIV patients are diagnosed. The centers will be selected based on the high proportion of patients at high risk visiting the EDs.

During targeted period, nurses will offer screening to all patients at EDs, aged 18-64 years old, identified as high-risk by a self-administered questionnaire, not know to be HIV positive, not being seen for post-exposure prophylaxis or unstable medical illness, and accepting to participate by providing an informed consent. The questionnaire was previously tested in one ED.

In case of reactive rapid test result, blood specimen will be collected for standard enzyme-linked immunosorbent assay and western blot confirmation. A follow-up visit with an on-site infectious disease specialist will be arranged within the following 48 hours.

Perspective :

This project will allow defining the benefit of nurse-driven HIV targeted screening in EDs and its potential utility to improve HIV screening in France.

ELIGIBILITY:
Inclusion Criteria:

* Patients at EDs, aged 18-64 years old and not being seen at ED for post exposure prophylaxis

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148327 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with newly identified HIV infection among the number of 18-64 years patients visited EDs (apart from being seen at ED for prophylaxis after exposure to HIV) during the inclusion periods | At the end of the expected total duration of the inclusion periods : up to 9 months in each center

SECONDARY OUTCOMES:
Linkage into care of patients with newly diagnosed infection (Follow-up visit with an on-site infectious disease specialist) | In the 3 months after the HIV screening at the emergency department
Number of new HIV positive tests among the total number of tests | At the end of the expected total duration of the inclusion periods : up to 9 months in each center
Early detection of HIV (Proportion of patients with CD4>500/mm3, >350/mm3 and >200/mm3, and without HIV-related symptoms at presentation) | In the 3 months after the HIV screening at the emergency department
Feasibility of the nurse-driven HIV screening (Proportion of : filled-questionnaires, proposition of the nurse-driven HIV screening, acceptation by patients and HIV rapid tests done by nurses) | At the end of the expected total duration of the inclusion periods : up to 9 months in each center
Acceptability of the nurse-driven HIV screening by the caregivers (Interviews with nurses, nurse managers, physician doctors and hospital managers) | Before and after the expected total duration of the inclusion periods : up to 9 months in each center
Cost-effectiveness of the 2 compared strategies | At the end of the expected total duration of the inclusion periods : up to 9 months in each center
Acceptability of the nurse-driven HIV screening by the patients (additional questionnaire proposed to patients in 4 centers) | Questionnaire proposed at ED for each patient after the main study questionnaire during inclusion period. Analysis after the expected total duration of the inclusion periods : up to 9 months in each center

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center (Centre de Recherche Clinique de l'Est Parisien, CRC-Est), Groupe Hospitalier des Hôpitaux Universitaires Est Parisien, Assistance Publique - Hôpitaux de Paris (AP-HP), Paris, France

REFERENCES:
- [Derived] Leblanc J, Hejblum G, Costagliola D, Durand-Zaleski I, Lert F, de Truchis P, Verbeke G, Rousseau A, Piquet H, Simon F, Pateron D, Simon T, Cremieux AC; DICI-VIH (Depistage Infirmier CIble du VIH) Group. Targeted HIV Screening in Eight Emergency Departments: The DICI-VIH Cluster-Randomized Two-Period Crossover Trial. Ann Emerg Med. 2018 Jul;72(1):41-53.e9. doi: 10.1016/j.annemergmed.2017.09.011. Epub 2017 Oct 31. PMID 29092761
- [Derived] Leblanc J, Rousseau A, Hejblum G, Durand-Zaleski I, de Truchis P, Lert F, Costagliola D, Simon T, Cremieux AC. The impact of nurse-driven targeted HIV screening in 8 emergency departments: study protocol for the DICI-VIH cluster-randomized two-period crossover trial. BMC Infect Dis. 2016 Feb 1;16:51. doi: 10.1186/s12879-016-1377-6. PMID 26831332